CLINICAL TRIAL: NCT00192751
Title: Impact of Psycho-Educational Intervention on Patients With Severe Mental Illness Recently Discharged From Psychiatric Inpatient Services
Brief Title: From Compliance to Alliance: Engaging Psychiatric Patients in Illness Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: compliance_CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-10-27 (Estimated); Status verified 2005-09

CONDITIONS: Patients Diagnosed With Severe Mental Illness
Keywords: Schizophrenia; Major depression; Bipolar disorder; Compliance; Relapse prevention
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder; Patient Compliance

INTERVENTIONS:
Behavioral: Psychoeducational group sessions

SUMMARY:
The purpose of this study is to determine the benefit and impact on relapse prevention,adherence to treatment and general health indices of participation in psycho-eduational group intervention among psychiatric patients with severe mental illness,recently discharged from inpatient services.

DETAILED DESCRIPTION:
Medication non-compliance, estimated to affect 50% of all psychiatric patients, was shown to be strongly associated with an elevated risk for relapse, readmission to psychiatric inpatient care, longer length of stay and suicide, resulting in elevated costs across the health care system. The proposed project seeks to bridge the gap between the significant progress of recent years in psycho-pharmacology that produced more efficient 'newer generation' medications, and the continuing unanswered problem of non-compliance, by applying knowledge from clinical decision-making theories and recent evidence-based research on the management of severe mental illness.

In Phase I of the project, an epidemiological survey will be conducted to evaluate the magnitude and correlates of the problem in patients attending walk-in crisis clinic , using Treatment Compliance Assessment and Decision-Making Assessment Tools, both developed by the researchers. An 8-module psycho-educational intervention protocol emphasizing illness management and optimization of health care decision-making will then be designed and implemented.

In Phase II, eligible outpatient clients will be randomly assigned to either Intervention or Standard Care conditions, and followed for a period of 15 months. Repeated assessments will include pre-post measures of knowledge, treatment compliance, and decision-making, and on outcome measures of relapse such as hospitalizations and symptoms, functioning, self-efficacy, quality of life, and satisfaction with services.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of severe mental illness, younger than 70 years of age, recently discharged from psychiatric inpatient services at the Rambam Medical Health Center.

Exclusion Criteria:

Diagnoses other than schizophrenia, major depression and bipolar disorders; 70 + years of age; organic problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-02; Study Completion 2006-12

PRIMARY OUTCOMES:
Relapse prevention
Illness management

SECONDARY OUTCOMES:
Satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Yael Caspi, Sc.D., M.A., Principal Investigator — Department of Psychiatry, Rambam Medical Center; Ehud Klein, MD, Study Chair — Department of Psychiatry, Rambam Health Center
Locations (1):
- Department of Psychiatry, Rambam Medical Center, Haifa, Israel